CLINICAL TRIAL: NCT04150471
Title: An Open Label, Observational Clinical Study to Assess Long-term Feasibility of Reduced Dose Dasatinib in Chronic Phase Chronic Myeloid Leukemia Patients Who Have Any Grade of Adverse Events and Early Molecular Response Within 3 Months of Frontline Dasatinib Therapy
Brief Title: Assess Long-term Feasibility of Reduced Dose Dasatinib in Chronic Phase Chronic Myeloid Leukemia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Dong-Wook Kim, Director, Seoul St. Mary's Hospital
Other Study IDs: DAS-CHANGE
Record Dates: First submitted 2019-10-20; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Chronic Myelocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Rest of RNA samples after Q-RT-PCR (Quantitative Real-time Polymerase chain reaction) analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: RQ-PCR(Real-time Quantitative Polymerase chain reaction) RNA Analysis — Conventional Q-RT-PCR every 3 months

SUMMARY:
This study is conducted in patients with newly diagnosed CP CML (Chronic Phase Chronic Myeloid Leukemia) who have achieved EMR (< 10% IS BCR-ABL) at 3 months after first line treatment with dasatinib. Subjects will be allocated to 80mg QD based on EMR (Early Molecular Response) achievement and early safety profile following a standard of care approach.

DETAILED DESCRIPTION:
Patients will sign the consent forms for screening prior to frontline dasatinib therapy (1st) and the 3 month molecular test date (2nd). The molecular samples will be analyzed in the central lab as part of the screening procedure.

Subjects will be treated for a maximum of 60 months after allocation of the last subject on the assigned regimen (dasatinib 80mg QD), unless disease progression, treatment failure or unacceptable toxicity occurs, the subject withdraws consent, or the study is discontinued by the sponsor. Subjects who discontinue study therapy early due to disease progression or intolerance to study medication will continue to be followed yearly for survival for up to 5 years after allocation of the last subject. All subjects will be followed yearly for progression-free survival and overall survival.

For patients who continue their assigned treatment, safety assessments will be conducted every 6 months and cytogenetic assessment as investigator assessment.

Follow up visits after the last dose of study drug will be required at least every 4 weeks until all study related toxicities resolve to baseline (or CTC Grade ≤ 1), stabilize or are deemed irreversible.

ELIGIBILITY:
Inclusion Criteria:

* Adult CML-CP Ph+ (Philadelpia) patients with BCR-ABL1 patients diagnosed within 3 months
* Adequate renal function defined as serum creatinine ≤ 3 times the institutional ULN(Upper limit of normal)
* Adequate hepatic function defined as: total bilirubin ≤ 2 times the institutional ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the institutional upper limit of normal (ULN).
* Adequate cardiac function (see exclusion criteria)
* Adequate pulmonary function (see exclusion criteria)
* Serum Na, K, Mg, and total serum Ca or ionized Ca levels must be greater than or equal to the institutional lower limit of normal. Subjects with low K, Mg levels, total serum Ca and/or ionized Ca must be replete to allow for protocol entry: Rescreening is permitted in the event of temporary biochemical abnormalities
* CML-CP Ph+ patients with CHR but with BCR-ABL level < 10% IS after 3 months of frontline dasatinib 100 mg treatment. And currently persisting any grade adverse events to dasatinib 100 mg QD
* ECOG(Eastern Cooperative Oncology Group) performance status 0-2
* Women must not be pregnant

Exclusion Criteria:

* Previous diagnosis of accelerated phase or blast crisis
* Documented any major ABL1 mutation
* A serious uncontrolled medical disorder or active infection that would impair the ability of the subject to receive dasatinib
* Pulmonary arterial hypertension
* Congenital bleeding disorders
* Prior or concurrent malignancy, except for the following
* Subject with any anti-CML other than dasatinib
* Subjects with prior stem cell transplantation and/or high dose chemotherapy for CML
* Subjects currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes
* Subjects who were previously treated with over 100mg at second phase screening
* Subjects who are not tolerable to 80mg at second phase screening
* Patients who are pregnant or breast feeding or likely to become pregnant
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult CML-CP Ph+ patients with BCR-ABL1 will start frontline dasatinib 100mg QD treatment. Dasatinib monotherapy must have been started within 3 months of CP-CML diagnosis. Patients having BCR-ABL1 transcript level < 10% IS (International Standard) after 3 months of treatment with frontline dasatinib will reduce dasatinib dose to 80mg QD and all of patients must have any grade of adverse events at 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of MMR | 12 month
  Level of Bcr-Abl transcript (Conventional Q-RT-PCR)

SECONDARY OUTCOMES:
To assess: Number and percentage of participants with treatment-related adverse events as assessed by CTCAE v4.0. | 12 months
  Safety
MMR and MR4.5 rates by 5 years | 5 years
  Level of Bcr-Abl transcript (Conventional Q-RT-PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Sahee Park, Study Director — Cancer Research Institute, The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cortes JE, Saglio G, Kantarjian HM, Baccarani M, Mayer J, Boque C, Shah NP, Chuah C, Casanova L, Bradley-Garelik B, Manos G, Hochhaus A. Final 5-Year Study Results of DASISION: The Dasatinib Versus Imatinib Study in Treatment-Naive Chronic Myeloid Leukemia Patients Trial. J Clin Oncol. 2016 Jul 10;34(20):2333-40. doi: 10.1200/JCO.2015.64.8899. Epub 2016 May 23. PMID 27217448